CLINICAL TRIAL: NCT07014670
Title: Validity and Reliability of the Postural Habits and Awareness Scale in Patients Diagnosed With Fibromyalgia in Turkey
Brief Title: Validity and Reliability of the Postural Habits and Awareness Scale
Status: Completed | Type: Observational
Sponsor: Bitlis Eren University (Other)
Responsible Party: Principal Investigator, Abdurrahman Tanhan, Research Assistant, Bitlis Eren University
Other Study IDs: BitlisErenU3
Record Dates: First submitted 2025-06-03; First posted 2025-06-11 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Fibromyalgia
Keywords: reability; validity; Postural Habit and Awareness Scale
MeSH Terms: conditions — Fibromyalgia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 3 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: Validation and Reability study — Validation and Reability study

SUMMARY:
The aim of this study was to examine the validity and reliability of the Turkish version of the Postural Habits and Awareness Scale in Fibromyalgia patients.

DETAILED DESCRIPTION:
Postural Habit and Awareness Scale is a scale developed for healthy individuals. For this reason, when applying to any disease group, other parameters belonging to that disease group should also be evaluated. For this purpose, Fibromyalgia Impact Questionnaire, Body Perception Scale, Body Awareness Questionnaire, Visual Analog Scale and Short Form-12 questionnaires were also used in the study. Fibromyalgia is a disease that affects the whole body and generally causes pain and stiffness complaints. For this reason, the whole body should be evaluated. Fibromyalgia Impact Questionnaire was used to define and indicate the level of fibromyalgia effects of the patients. For validity and reliability analyses, Body Perception Scale and Body Awareness Questionnaire questionnaires were used to compare the Postural Habit and Awareness scale. At the same time, Short Form-12 questionnaire was used to examine the patients' pain severity and the effects of the disease on daily life.

ELIGIBILITY:
Inclusion Criteria:

* Those who have been diagnosed with Fibromyalgia according to the American Rheumatology Association criteria and have been over for at least 6 months,
* Those who do not have a history of any psychiatric disease,
* Those who have the ability to lie down, sit and stand without any assistance.

Exclusion Criteria:

* Pregnant individuals,
* Those who have pain complaints due to another disease (rheumatic, heart or infectious diseases),
* Those who make changes in physical activity and lifestyle during work,
* Those with any neurological disease

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Fibromyalgia
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-04-25 (Actual); Primary Completion 2025-06-30 (Actual); Study Completion 2025-06-30 (Actual)

PRIMARY OUTCOMES:
Postural Habit and Awareness Scale | 7-10 days
  Developed by Turkish researchers Bayar and his colleagues, the scale has 19 items and four factors. The factors of the scale are posture habits and awareness, awareness of factors that disrupt posture, positional awareness and ergonomic awareness. Postural habits are examined with seven items and postural awareness is examined with twelve items in the scale. Scoring is 5-point Likert type, the minimum score is one for each proposition; the maximum score is five. The total score is a maximum of 95.

SECONDARY OUTCOMES:
Fibromyalgia Impact Questionnaire | 2 days
  The questionnaire consists of 10 propositions. It is a tool that allows the patient to evaluate themselves in terms of physical function, work status, depression, anxiety, sleep, pain, stiffness, fatigue and feeling good. The questionnaire has a 4-point Likert structure and the scoring varies between 0-3. A high score means that physical disability increases
Body Perception Scale | 2 days
  It is a tool that allows the patient to evaluate their body perception themselves. It consists of 46 items in total. The scale is scored between 1-5, with a high score indicating poor body image.
Body Awareness Questionnaire | 2 days
  This questionnaire is designed to determine the normal and/or abnormal sensitivity level of an individual's body composition. This questionnaire consists of four subgroups. These subgroups are; changes in body processes, sleep-wake cycle, prediction at the beginning of the disease, prediction of body reactions. BFA is a 7-point Likert type scale and consists of 18 items in total. Each item is scored between 1-7. The lowest possible score is 18, and the highest score is 126
Visual Analog Scale | 2 days
  VAS is a reliable and easily applicable scale that is accepted in the literature and used to measure the pain intensity of patients. The patient is asked to mark the part that represents the pain intensity on a straight line between 0-10 cm. The "0" at the beginning indicates no pain, and the "10" at the end indicates the presence of very severe, unbearable pain
Short Form-12 | 2 days
  This form; It consists of 8 sub-dimensions and 12 items: physical functioning, physical role, body pain, general health, energy, social functioning, emotional role and mental health. The Physical Component Summary and Mental Component Summary scores of the scale are calculated separately. The Physical Component Summary -12 score is obtained from the general health, physical functioning, physical role and body pain sub-dimensions. The Mental Component Summary -12 score is scored with the social functioning, emotional role, mental health and energy sub-dimensions. The scores of both sub-dimensions vary between 0-100. A higher score indicates a better quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Bitlis Eren University, Bitlis, Merkez, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No